CLINICAL TRIAL: NCT07331883
Title: Sintilimab Combined With Bevacizumab Biosimilar as Adjuvant Treatment After Resection of Ruptured Hepatocellular Carcinoma: A Prospective, Exploratory, Single-Arm Study (CLEAR-2)
Brief Title: Sintilimab Combined With Bevacizumab Biosimilar as Adjuvant Treatment After Resection of Ruptured Hepatocellular Carcinoma (CLEAR-2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR-2
Record Dates: First submitted 2025-11-26; First posted 2026-01-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Sintilimab (200 mg, iv, d1, q3w) in combination with bevacizumab biosimilar (15mg/kg, iv, d1, q3w)
  Interventions: Drug: Sintilimab plus bevacizumab biosimilar

INTERVENTIONS:
Drug: Sintilimab plus bevacizumab biosimilar — Sintilimab (200 mg, iv, d1, q3w) in combination with bevacizumab biosimilar (15mg/kg, iv, d1, q3w)

SUMMARY:
Primary liver cancer-particularly hepatocellular carcinoma (HCC)-remains a major health burden in China, characterized by high incidence and mortality rates and poor 5-year survival. Spontaneous rupture of HCC (SRHCC), although a relatively uncommon complication, is associated with extremely high mortality and marked geographic variation, with disproportionately higher incidence and rupture-related deaths reported in Asian populations. For patients with preserved liver function and resectable tumors, hepatic resection can offer favorable long-term survival and even a potential cure. However, despite surgical removal, the risk of postoperative recurrence is substantially increased, and long-term outcomes remain unsatisfactory. Currently, there is no validated adjuvant therapy to reduce recurrence or improve survival after resection.

In recent years, immune checkpoint inhibitors (ICIs) in combination with anti-angiogenic agents have demonstrated synergistic antitumor activity and manageable safety in advanced HCC. Notably, studies of sintilimab plus a bevacizumab biosimilar have shown significant improvements in overall survival (OS), progression-free survival (PFS), and objective response rate (ORR). Moreover, emerging evidence in the adjuvant and perioperative settings suggests that PD-1 blockade may delay recurrence in high-risk patients, such as those with microvascular invasion.

Based on the high postoperative recurrence rate in SRHCC patients and the existing therapeutic gap, along with established evidence of the efficacy of immune checkpoint inhibitors combined with antiangiogenic therapy in advanced HCC, conducting a prospective Phase II single-arm study of adjuvant therapy with sintilimab plus the bevacizumab biosimilar holds significant clinical and scientific value. This study aims to evaluate the tolerability of this combination regimen in postoperative SRHCC patients at high risk of recurrence. It is expected to provide a more effective treatment option for patients diagnosed with spontaneously ruptured hepatocellular carcinoma, improve their prognosis, and offer scientific evidence for future treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily provide written informed consent, with authorization obtained from the patient or legal representative prior to any protocol-related procedures.
* Age ≥ 18 years and ≤ 75 years; both female and male
* Spontaneous tumor rupture with hemorrhage confirmed by imaging prior to or during surgery, with a postoperative pathological diagnosis of hepatocellular carcinoma (HCC).

  a) For cases where tumor rupture is an incidental finding during surgery, a clinical history of abdominal pain within the two weeks preceding surgery is required.
* CNLC Stage I-II.
* Having undergone curative surgical resection, with intraoperative irrigation using ≥5000 mL of distilled water or normal saline, confirmed negative surgical margins on postoperative pathology, and achieving a complete response (CR) confirmed by imaging within 4-8 weeks after surgery.
* ECOG PS 0-1
* Child-Pugh A (score ≤6).
* Life expectancy ≥12 months
* Laboratory test results obtained within 3 days prior to the first dose must meet the following criteria:

  1. Hematological:(Except for hemoglobin, the patient must not have received a blood transfusion, granulocyte colony-stimulating factor [G-CSF], or hematopoietic agents within 2 weeks prior to screening.) i. Absolute neutrophil count ≥1.5 × 10⁹/L; ii. Platelet count ≥75 × 10⁹/L; iii. Hemoglobin ≥90 g/L.
  2. Serum biochemistry:

     i. Serum albumin ≥30 g/L; ii. Total bilirubin ≤1.5 × ULN; iii. ALT and AST ≤3 × ULN; iv. Serum creatinine ≤1.5 × ULN, or creatinine clearance >50 mL/min.
  3. International normalized ratio (INR) ≤1.2 or prothrombin time (PT) ≤2 seconds above the upper limit of normal.
  4. Urinalysis:Urine protein <2+.(If urine protein is ≥2+, a 24-hour urine protein test may be performed; patients may be enrolled if 24-hour urine protein <1.0 g.)
* For patients with HBV infection (i.e., HBsAg-positive), HBV DNA must be tested. HBV DNA levels must be <2000 IU/mL (or <10⁴ copies/mL if the study site reports results in copies/mL). Patients with HBV DNA ≥2000 IU/mL must receive at least 1 week of antiviral therapy prior to the first dose, using only nucleos(t)ide analogues such as entecavir, tenofovir disoproxil fumarate, or tenofovir alafenamide. HBV DNA levels must show a ≥1-log (10-fold) reduction before initiation of study treatment. All HBV-infected patients must continue antiviral therapy throughout the entire study period. Patients who are HCV RNA-positive must receive antiviral treatment according to current clinical guidelines.
* Female patients of childbearing potential must have a negative β-hCG pregnancy test prior to the first dose. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use effective contraception during treatment and for 6 months after the last dose of study medication.

Exclusion Criteria:

* Pathological diagnosis other than hepatocellular carcinoma, including cholangiocarcinoma or combined hepatocellular-cholangiocarcinoma.
* Intraoperative intraperitoneal lavage with chemotherapeutic agents
* Child-Pugh class B or C
* ECOG PS > 1
* Postoperative imaging confirming the presence of extrahepatic metastasis, residual disease, or recurrence.
* Prior systemic antitumor therapy, including targeted therapy, immunotherapy, investigational drugs, or local therapies such as TACE (preoperative TAE for hemostasis is allowed). Patients who received adjuvant TACE after resection are also excluded.
* Clinically symptomatic moderate or severe ascites requiring therapeutic paracentesis or drainage, or a Child-Pugh ascites score >2 (the presence of minimal ascites on imaging only, without associated symptoms, is excluded). Uncontrolled or moderate-to-large pleural effusion or pericardial effusion.
* Current interstitial lung disease (ILD), or a history of ILD requiring glucocorticoid treatment, or other conditions that might interfere with the diagnosis or management of immune-related pulmonary toxicity, including pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), pneumoconiosis, drug-induced pneumonia, or idiopathic pneumonia. Patients with evidence of active pneumonia on screening chest computed tomography (CT) scans or severely impaired pulmonary function are excluded. History of radiation pneumonitis within the radiation field is permitted. Active tuberculosis.
* Presence of an active autoimmune disease, or a history of autoimmune disease with potential for recurrence [including, but not limited to, autoimmune hepatitis, pneumonitis, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients with hypothyroidism controlled only with hormone replacement therapy are eligible)]. Patients with vitiligo, psoriasis, or alopecia not requiring systemic treatment, or well-controlled type I diabetes on insulin, or childhood asthma that has completely resolved in adulthood without any intervention are eligible. Asthmatic patients requiring bronchodilators for medical intervention are excluded.
* Use of immunosuppressive agents or systemic corticosteroids for immunosuppressive purposes (at doses >10 mg/day prednisone or equivalent) within 2 weeks prior to initiation of study treatment. Inhaled or topical corticosteroids, and adrenal replacement steroid doses ≤10 mg/day prednisone equivalent, are permitted in the absence of active autoimmune disease.
* History of gastrointestinal bleeding within 6 months prior to treatment, or definite predisposition to gastrointestinal bleeding, such as high-risk or severe esophageal/gastric varices, active peptic ulcer disease, or persistently positive fecal occult blood test (unless follow-up endoscopy rules out high-risk varices). Patients with esophageal/gastric varices identified on baseline CT/MRI may be eligible if assessed by the investigator as mild to moderate. Presence of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to randomization.
* Known hereditary or acquired bleeding (e.g., coagulation disorders) or thrombotic tendency, such as hemophilia, coagulopathy, thrombocytopenia, etc. Current therapeutic use of full-dose oral or injectable anticoagulants or thrombolytic agents (prophylactic use of low-dose aspirin, etc., is permitted).
* History of thrombotic or embolic events within 6 months prior to treatment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
* Poorly controlled or significant cardiac disease, including: (1) Cardiac dysfunction ≥ Grade II per New York Heart Association (NYHA) classification, or left ventricular ejection fraction (LVEF) <50% on echocardiography; (2) Unstable angina; (3) Myocardial infarction within 1 year prior to initiation of study treatment; (4) Clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) QTc interval >450 ms (males) or >470 ms (females).
* Hypertension that is not adequately controlled with antihypertensive medication (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, based on the average of ≥2 readings). History of hypertensive crisis or hypertensive encephalopathy.
* Major vascular disease within 6 months prior to treatment (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis).
* Severe, non-healing, or dehisced wounds, active ulcers, or unhealed bone fractures.
* Inability to swallow tablets, malabsorption syndrome, or any condition compromising gastrointestinal absorption.
* Severe infection within 4 weeks prior to treatment, including, but not limited to, hospitalization for infection, bacteremia, or severe pneumonic complications. Therapeutic antibiotics (oral or intravenous) within 14 days prior to randomization (prophylactic antibiotic use is permitted). Unexplained fever ≥38.5°C within 7 days prior to randomization, or baseline white blood cell count >15×10⁹/L.
* Known congenital or acquired immunodeficiency (e.g., HIV infection).
* Administration of live attenuated vaccines within 28 days prior to treatment, or anticipation of need for such vaccines during the study period.
* Any other condition that, in the investigator's judgment, may affect the interpretation of results, compromise patient safety, or lead to premature study termination. This includes alcohol or substance abuse, other severe concurrent illnesses (including psychiatric disorders) requiring treatment, severe laboratory abnormalities, or significant social/familial circumstances.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
DIsease-free Survival (DFS) | Through out the study (up to 3 years)
  The time from initial curative-intent treatment to the date of the first documented tumor progression as determined by the investigator (per RECIST 1.1), or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Through out the study (up to 3 years)
  the time from initial curative-intent treatment until death due to any cause.
Adverse Event description as assessed by CTCAE V5.0 | Through out the study (up to 3 years)
  Number of Participants With Abnormal Laboratory Values and Adverse Events That Are Related to Treatment
the proportion and timing of intrahepatic recurrence | Through out the study (up to 3 years)
  documenting the proportion and timing of intrahepatic recurrence
the proportion and timing of extrahepatic metastasis | Through out the study (up to 3 years)
  the proportion and timing of extrahepatic metastasis
the proportion and timing of peritoneal metastasis | Through out the study (up to 3 years)
  the proportion and timing of peritoneal metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No